CLINICAL TRIAL: NCT07001436
Title: A Non-randomized, Open, Parallel, Single-dose Pharmacokinetics and Safety Study of Azvudine Tablets in Subjects With Mild-To-Moderate GFR Decline in Renal Insufficiency and in Healthy Subjects
Brief Title: A Pharmacokinetics and Safety Study of Azvudine Tablets in Subjects With Mild-To-Moderate GFR Decline in Renal Insufficiency and in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-FNC-RI-102
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Renal Insufficiency
Keywords: Azvudine
MeSH Terms: conditions — Renal Insufficiency | interventions — azvudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : subjects with mildly decreased GFR(GRF, Glomerular Filtration Rate) (Experimental)
  Interventions: Drug: Azvudine tablets
- Group 2 : subjects with a moderate decrease in GFR (Experimental)
  Interventions: Drug: Azvudine tablets
- Group 3 : healthy subjects matched with group 1 and group 2 (Experimental)
  Interventions: Drug: Azvudine tablets

INTERVENTIONS:
Drug: Azvudine tablets — On the first day of the study, a single oral dose of 3 mg ( 3 tablets ) of Azvudine tablets is taken orally on an empty stomach.

SUMMARY:
Azvudine(FNC)，a nucleoside reverse transcriptase inhibitor, make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance. FNC is a broad-spectrum RNA virus inhibitor that inhibits the novel coronavirus RNA-dependent RNA polymerase.

This trial uses a non-randomized, open-label, parallel, single-dose adaptive design aimed at investigating the effects of varying degrees of renal insufficiency on the pharmacokinetics, safety, and tolerability of a single oral dose of 3 mg Azvudine tablets in humans. On the first day of the study, a single oral dose of 3 mg ( 3 tablets ) of Azvudine tablets is taken orally on an empty stomach. Biological sample collection and safety examination will be performed in this trial.

ELIGIBILITY:
Inclusion Criteria:

(一) Renal insufficiency study participants and healthy study participants:

1. Age ≥ 18 years old and ≤ 70 years old, regardless of gender;
2. Body mass index (BMI) within the range of 18.0-30.0 (including the critical value) (BMI = weight (kg) / height 2 (m2)), the weight of men should be ≥ 50.0kg, and the weight of women should be ≥ 45.0kg;
3. Females of childbearing potential must have taken reliable and highly effective contraceptive measures and have a negative baseline blood pregnancy test at screening, and are willing to use appropriate and efficient methods of contraception after signing the informed consent form until 3 months after the last dose of the test drug; Male study participants who are willing to do so for the duration of the trial and for 3 months after the last dose of the trial drug Have no plans to have children and voluntarily use highly effective contraception, or have been surgically sterilized;
4. Understand and sign the informed consent form.

(二) Health study participants (in addition to the above criteria, they should also meet):

1. The health condition is judged by the investigator to be good, and the results of vital signs, physical examination, electrocardiogram, and laboratory examination are normal or abnormal, and there is no clinical significance;
2. Those who have not taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health care products within 14 days before screening;
3. Meet the classification standard of glomerular filtration rate of 90≤GFR<130 ml/min;
4. Study participants with mild or moderate decline in GFR were matched with the following demographic characteristics: age (mean ± 10 years), weight (mean ±10kg), and gender (±1 cases).

(三) Renal insufficiency study participants (in addition to the above criteria, they should also meet):

1. Stable renal function status: the existing renal function impairment is required to last for more than 3 months, and the GFR results of two tests (with an interval of 72 hours or more) during the screening period are within the same grade and the difference between the two tests is not more than 25%;
2. No clinically significant abnormalities were found in the pre-test medical history, vital signs, physical examination, laboratory test items (except ALT and AST, total bilirubin, and direct bilirubin) and test-related examinations and were judged by the clinical research physician to be eligible for enrollment (except for abnormalities related to renal impairment);
3. The drug being taken by the study participant with renal insufficiency, which should not affect the absorption, distribution, metabolism or excretion of the study drug, and has been taken at a stable dose for at least 4 consecutive weeks before giving the study drug, and agrees to continue treatment during the study period;
4. Two weeks before administration and during the test, Chinese patent medicines, traditional Chinese medicine decoctions, ethnic medicines, SGLT-2i, MRA drugs and benzbromarone are prohibited;
5. During the screening period, it is necessary to meet: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), and direct bilirubin (DBIL) all need to < 1.5 upper limit of normal (ULN)
6. Participants in the study of renal insufficiency of all grades met the grading criteria for glomerular filtration rate (GFR was taken as the average of the two tests during the screening period): Mild decrease in GFR: 60≤ GFR≤89 ml/min; Moderate decrease in GFR: 30≤GFR ≤59 ml/min.

Exclusion Criteria:

(一) Renal insufficiency and health research participants:

1. Allergies, especially those who are allergic to any of the ingredients in this product and excipients;
2. Those who have undergone gastrointestinal resection in the past, or suffer from digestive diseases that will affect the absorption, distribution, metabolism and excretion of drugs;
3. Those who have a history of drug abuse within 12 months before screening or those who have tested positive for addictive substances before enrollment;
4. Those with fever or infectious diseases at the time of screening;
5. Those who have participated in other clinical trials within 3 months before screening;
6. Those who have a history of smoking addiction within 12 months before screening (the average number of cigarettes per day ≥5);
7. Those who have a history of alcohol abuse within 12 months before screening (drinking ≥ 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 150mL of wine) or positive alcohol breath test (test value >0mg/100mL) before enrollment;
8. Those who have lost blood or donated 200mL of blood ≥ within 8 weeks before screening;
9. Hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, treponema pallidum antibody or rapid plasma reagin ring card test (RPR) test results are positive.
10. Pregnant and lactating women;
11. Those who cannot tolerate vascular puncture blood collection and/or have a history of blood sickness, needle fainting and/or poor blood collection vascular conditions;
12. Those who have been vaccinated within 3 months before screening, or plan to be vaccinated during the trial;
13. Those who are not considered suitable to enter this trial by the investigator.

(二) Renal insufficiency study participants (except for the above criteria):

1. Have undergone kidney transplantation;
2. Systolic blood pressure outside the range of 90 ~ 160mmHg, diastolic blood pressure outside the range of 50 ~ 100mmHg, or heart rate outside the range of 50 ~ 120bpm;
3. Frequent occurrence of hypoglycemia and exclusion of drug factors within 3 months prior to screening;
4. Albumin<30g/L;
5. Hemoglobin value<9 g/dL;
6. Those who have a history of uncontrolled or unstable serious diseases of cardiovascular, liver, pulmonary, digestive tract, nerves, autoimmune, metabolic and musculoskeletal systems, hematopoietic systems and other systems, or those whose diseases are active.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Azvudine | Blood samples: up to 48 hours post-dose; urine samples：up to 72 hours post-dose
  Cmax will be calculated by measuring the concentration of Azvudine in blood samples and urine samples.
Pharmacokinetics (PK): Area Under the Concentration-Time Curve from the First Dose to the Last Blood Collection Point (AUC0-t) of Azvudine | Blood samples: up to 48 hours post-dose; urine samples：up to 72 hours post-dose
  AUC0-t will be calculated by measuring the concentration of Azvudine in blood samples and urine samples.
Pharmacokinetics (PK): Area Under the Concentration-Time Curve Extrapolated from the Initial Administration to Infinity (AUC0-∞) of Azvudine (if applicable) | Blood samples: up to 48 hours post-dose; urine samples：up to 72 hours post-dose
  AUC0-∞ will be calculated by measuring the concentration of Azvudine in blood samples and urine samples.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of Azvudine | Blood samples: up to 48 hours post-dose; urine samples：up to 72 hours post-dose
  Tmax will be calculated by measuring the concentration of Azvudine in blood samples and urine samples.
Pharmacokinetics (PK): Elimination Half-life (t1/2) of Azvudine | Blood samples: up to 48 hours post-dose; urine samples：up to 72 hours post-dose
  t1/2 will be calculated by measuring the concentration of Azvudine in blood samples and urine samples.
Occurrence of Adverse Events | From enrollment to the end of the study on Day 4.
  Clinical presentation characteristics, severity, onset time, duration of adverse events, management measures, outcomes, and the correlation with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China